CLINICAL TRIAL: NCT05757973
Title: Pre-Approval Access Named Patient Program for Talquetamab (JNJ-64407564) for Treating Physician Use in Relapsed or Refractory Multiple Myeloma
Brief Title: Pre-Approval Access Program for Talquetamab in Relapsed or Refractory Multiple Myeloma
Status: Approved for marketing | Type: Expanded Access
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: CR109170; 64407564MMY4003 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2022-12-14; First posted 2023-03-07 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — talquetamab

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Talquetamab — Talquetamab will be administered subcutaneously.
  Other Names: JNJ-64407564

SUMMARY:
The purpose of this pre-approval access program is to give talquetamab monotherapy (treatment with single drug) to participants with relapsed or refractory multiple myeloma (a type of cancer that begins in plasma cells [white blood cells that produce antibodies] which has returned or difficult to treat) who have relapsed on or are refractory to all locally available and clinically appropriate treatment and who are not eligible for a clinical trial.

DETAILED DESCRIPTION:
Talquetamab (JNJ-64407564) is a humanized immunoglobulin G4 proline, alanine, alanine (IgG4PAA) bispecific antibody designed to target G-Protein Coupled Receptor (5DGPRC5D) and cluster of differentiation 3 (CD3). Redirecting T-cells to a tumor surface antigen using bispecific antibody approaches may be an effective means to harness the immune system to destroy cancer cells expressing GPRC5D and create meaningful and long-lasting clinical responses. Talquetamab is supplied as single-dose Investigational Product (IP) vials for subcutaneous administration. Safety assessments will include adverse events, serious adverse events, adverse drug reactions, and special situations which will be reported during the duration of the pre-approval access program.

ELIGIBILITY:
Inclusion Criteria:

* Participant diagnosed with relapsed or refractory multiple, myeloma
* Participant exhausted all commercially approved and clinically appropriate treatment options, and is ineligible for a clinical trial

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC